CLINICAL TRIAL: NCT06977035
Title: Nerve Conduction Study for Assessment of Peripheral Neuropathy in Rheumatoid Arthritis Patients on the Janus Kinase Inhibitor Baricitinib
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Khairy Mohamed, Resident at Physical medicine, Rheumatology and Rehabilitation Department, Sohag University Hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh--Med--25-4-09MS
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Nerve Conduction Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rheumatoid Arthritis patients on Baricitinib treatment (Active Comparator)
  Interventions: Device: Nerve Conduction Study
- Rheumatoid Arthritis patient on conventional synthetic DMARD (Active Comparator)
  Interventions: Device: Nerve Conduction Study

INTERVENTIONS:
Device: Nerve Conduction Study — Sensory and Motor Nerve Conduction study on upper and lower limbs.

SUMMARY:
Rheumatoid arthritis is a chronic, systemic, autoimmune inflammatory disease that mainly affects the joints and periarticular soft tissues. Baricitinib (Olumiant®) is an oral, targeted synthetic DMARD that inhibits JAK1 and JAK2, which are implicated in the pathogenesis of rheumatoid arthritis (RA). Nerve conduction studies (NCSs) are an essential tool in the evaluation of the peripheral nervous system. The sensory nerve action potential (SNAP) provides information on the sensory nerve axon and its pathway from the distal receptors in the skin to the dorsal root ganglia, while the compound muscle action potential (CMAP) is an assessment of the motor nerve fibers from their origins in the anterior horn cell to their termination along muscle fibers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients fulfill the 2010 ACR/EULAR classification criteria of RA
2. Age above 18 years old.
3. Patient cooperative and can answer questions

Exclusion Criteria:

1. Other rheumatologic or collagen diseases.
2. Age below 18 years and above 65 years.
3. Uncooperative patients.
4. Patients with other causes of peripheral neuropathy as Diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
prevalence of Peripheral Neuropathy in Rheumatoid Arthritis Patients on Baricitinib | 6 months
  Assessment of Peripheral Neuropathy in Rheumatoid Arthritis Patients on Baricitinib in comparison to those on conventional synthetic DMARDs.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Di Matteo A, Bathon JM, Emery P. Rheumatoid arthritis. Lancet. 2023 Nov 25;402(10416):2019-2033. doi: 10.1016/S0140-6736(23)01525-8. Epub 2023 Oct 27. PMID 38240831
- [Background] Grassi W, De Angelis R, Lamanna G, Cervini C. The clinical features of rheumatoid arthritis. Eur J Radiol. 1998 May;27 Suppl 1:S18-24. doi: 10.1016/s0720-048x(98)00038-2. PMID 9652497
- [Background] Al-Salama ZT, Scott LJ. Baricitinib: A Review in Rheumatoid Arthritis. Drugs. 2018 May;78(7):761-772. doi: 10.1007/s40265-018-0908-4. PMID 29687421
- [Background] Mallik A, Weir AI. Nerve conduction studies: essentials and pitfalls in practice. J Neurol Neurosurg Psychiatry. 2005 Jun;76 Suppl 2(Suppl 2):ii23-31. doi: 10.1136/jnnp.2005.069138. No abstract available. PMID 15961865